CLINICAL TRIAL: NCT02626741
Title: Effect of a Meal Replacement on Weight Loss Obesity Patients With Metabolic Syndrome : A Randomized Controlled Trial
Brief Title: Effect of a Meal Replacement on Weight Loss Obesity Patients With Metabolic Syndrome
Acronym: SlimWell
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 647-2557-EC4
Record Dates: First submitted 2015-12-04; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Abdominal Obesity-Metabolic Syndrome
MeSH Terms: conditions — Abdominal obesity metabolic syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- meal replacement group (Experimental): the participants receive a meal replacement plus life style modification
  Interventions: Dietary Supplement: meal replacement group; Behavioral: control group
- control group (Experimental): the participants receive life style modification only.
  Interventions: Behavioral: control group

INTERVENTIONS:
Dietary Supplement: meal replacement group — The participants will receive SlimWell 60 grams per meal for 2 meals per day plus life style modification including educational sessions of exercise, dietary intake, food record. The duration is 3 months.
  Other Names: SlimWell
  Arms: meal replacement group
Behavioral: control group — The participants will receive only life style modification including educational sessions of exercise, dietary intake, food record. The duration is 3 months.
  Other Names: only life style modification

SUMMARY:
The purpose of this study is to determine whether meal replacement, SlimWell ®, is effective in the treatment of obesity patients with metabolic syndrome.

DETAILED DESCRIPTION:
The participants are divided into two groups: intervention group and control group. In the intervention group, the participants receive a meal replacement plus life style modification. In the control group, the participants receive only life style modification.

Sample size calculation is 69 participants per group. Primary outcome is to compare the weight loss between the intervention group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index more than or equal to 25 kg/m2
* Patients with metabolic syndrome
* Patients who are on anti-hypertensive drugs, oral hypoglycemic drugs and lipid lowering drugs.

Exclusion Criteria:

* Uncontrolled diabetes patients
* Patients with gastrointestinal abnormalities
* Patients with cardiovascular diseases
* Patients with hematologic disorders
* Patients with Glomerular filtration rate less than 60 ml/min/1.73m2
* Patients with drug or alcohol abuse
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Participants with weight loss unit in kilograms | 3 months
  Change from baseline body weight at 3 months

SECONDARY OUTCOMES:
Participants with waist circumference change in centimeters | 3 months
  Change from baseline waist circumference at 3 months
Participants with triglyceride change in mg/dl. | 3 months
  Change from baseline triglyceride at 3 months
Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study meal replacement, Graded According to NCI CTCAE Version 3.0 | 3 months
  Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study meal replacement, Graded According to NCI CTCAE Version 3.0 focus on Gastrointestinal side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Kusuma Chaiyasoot, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Leader NJ, Ryan L, Molyneaux L, Yue DK. How best to use partial meal replacement in managing overweight or obese patients with poorly controlled type 2 diabetes. Obesity (Silver Spring). 2013 Feb;21(2):251-3. doi: 10.1002/oby.20057. PMID 23404963